CLINICAL TRIAL: NCT05089877
Title: Outcomes of Surgical AF Ablation Using cryoICE Cryoablation System
Brief Title: FREEZE-AFIB Post-Market Study
Status: Completed | Type: Observational
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-2021-02
Record Dates: First submitted 2021-08-16; First posted 2021-10-22 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Surgical ablation; Cryo probe
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Surgical Ablation — The AtriCure cryoICE® cryoFORMTM cryoablation probe is used in the cryosurgical treatment of cardiac arrhythmias by freezing target tissues, creating an inflammatory response (cryonecrosis) that blocks the electrical conduction pathway.

SUMMARY:
This study is proposed herein is to gather clinical data on the safety and performance of the CRYOF device.

DETAILED DESCRIPTION:
This study is proposed herein is to gather clinical data on the safety and performance of the CRYOF device. Specifically, data from this study will be used for submission to regulatory authorities in Europe, China and other geographies as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than or equal to 18 years of age.
2. Subject has documented history of atrial fibrillation.
3. Subjects who received surgical ablation for their atrial fibrillation using CRYOF and on whom at least the following lesions were performed: Left and right pulmonary vein isolation, roof and floor lines, mitral annulus line and a connecting lesion from left atrial appendage to left pulmonary vein coronary sinus lesion and LAA exclusion , with a lesion duration of at least 2 minutes.
4. Stable subject that underwent non-emergent cardiac surgical procedure(s) on cardiopulmonary bypass including open-heart surgery for one or more of the following: mitral valve repair or replacement, aortic valve repair or replacement, tricuspid valve repair or replacement, or coronary artery bypass procedures, or atrial septal defect (ASD) repair
5. Left Ventricular Ejection Fraction ≥ 30% (determined by echocardiography or cardiac catheterization performed within 90 days of enrollment as documented in patient medical history).
6. Subject is willing and able to provide written informed consent.
7. Subject is willing and able to return for scheduled follow-up visits.

Exclusion Criteria:

1. Stand-alone AF without indication(s) for concomitant CABG and/or valve surgery.
2. Previous left sided ablation procedures procedure.
3. Untreated atrial flutter and symptomatic ventricular arrythmia
4. Known carotid artery stenosis greater than 80% prior to index ablation procedure.
5. Prior history of ischemic stroke or hemorrhagic stroke
6. History of MI with ST elevation within 6 weeks prior to the index ablation
7. Documented AF duration of greater than 10 years.
8. Large left atrial size i.e., LA diameter >7 cm prior to the index ablation procedure.
9. Subjects with active systemic infection prior to index ablation procedure.
10. Subjects who had documented severe peripheral arterial occlusive disease defined as claudication with minimal exertion prior to the ablation procedure.
11. Subjects with history of renal failure requiring dialysis or hepatic failure prior to the ablation procedure.
12. A known drug and/or alcohol addiction.
13. Mental impairment or other conditions which may not allow the subject to understand the nature, significance, and scope of the study.
14. Subjects who are pregnant
15. Subjects who had preoperative need for mechanical circulatory support or intravenous inotropes.
16. Subjects who are on anti-arrhythmic drug therapy for the treatment of another arrhythmia.
17. Subjects in currently undergoing chemotherapy.
18. Subjects on long term treatment with oral or injected steroids (not including intermittent use of inhaled steroids for respiratory diseases).
19. Subjects who had known connective tissue disorders at the time of index ablation procedure
20. Subjects who had known hypertrophic obstructive cardiomyopathy at the time of index ablation procedure
21. Subjects with known cold agglutinin.
22. Subjects who had or tested positive for COVID-19
23. Subjects with bleeding disorders and/or inability to receive anticoagulation
24. Subjects undergoing aortic dissection surgery as index procedure.
25. Cardiac surgical re-intervention since the index cardiac surgery with concomitant AF ablation procedure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone concomitant surgical AF ablation using the CRYOF device under investigation.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Hartford Hospital, Hartford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Northwestern University, Evanston, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Saint Thomas West Hospital, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Randomized, Single Arm Study: Patients who have undergone concomitant surgical AF ablation using the CRYOF device under investigation.
Period: Overall Study
Arm/Group | Non-Randomized, Single Arm Study
Started | 39
Completed | 28
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Non-Randomized, Single Arm Study
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants] — Population: Out of 39 participants, some participants were lost to follow up and some did not meet inclusion criteria.
  Participants
    number analyzed (Participants) | 33
    <=18 years | 0
    Between 18 and 65 years | 13
    >=65 years | 20
Age, Continuous [Mean (Full Range); unit: years] — Population: Out of 39 participants, some participants were lost to follow up and some did not meet inclusion criteria.
  years
    number analyzed (Participants) | 33
    (all) | 68.7 [53 to 83]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Out of 39 participants, some participants were lost to follow up and some did not meet inclusion criteria.
  Participants
    number analyzed (Participants) | 33
    Female | 8
    Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Out of 39 participants, some participants were lost to follow up and some did not meet inclusion criteria.
  Participants
    number analyzed (Participants) | 33
    Hispanic or Latino | 1
    Not Hispanic or Latino | 32
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Out of 39 participants, some participants were lost to follow up and some did not meet inclusion criteria.
  Participants
    number analyzed (Participants) | 33
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 31
    More than one race | 0
    Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Death, Stroke (Regardless of Level of Disability), Myocardial Infarction, and Major Bleeding Events.
Description: Death, stroke (regardless of level of disability), myocardial infarction, and major bleeding events within 30-days of the index ablation procedure. Measured by number of patients with Treatment-Related Adverse Events.
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Randomized, Single Arm Study
Number analyzed (Participants) | 33
Participants | 0

2. Primary Outcome: Freedom From Any Documented AF, AFL or AT Lasting >30 Seconds in the Duration of the Last Follow-up Visit Off Antiarrhythmic Therapy (Except of AADs at Doses Not Exceeding Those Previously Failed
Description: Freedom from any documented atrial fibrillation (AF), atrial flutter (AFL), or atrial tachycardia (AT) lasting >30 seconds in duration at the last follow-up visit off antiarrhythmic therapy (except of AADs at doses not exceeding those previously failed). Measured by 24-hour Holter Monitoring.
Time Frame: 12-24 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Randomized, Single Arm Study
Number analyzed (Participants) | 28
Participants | 25

3. Secondary Outcome: Freedom From Any Documented AF, AFL, or AT Lasting >30 Seconds at the Last Follow-up Visit Regardless of Class I or III AADs
Description: Freedom from any documented AF, AFL, or AT lasting >30 seconds at the last follow-up visit regardless of Class I or III AADs.
Time Frame: 12-24 months post procedure
Reporting Status: Not Posted

4. Secondary Outcome: Freedom From Any Documented AF, AFL, or AT Lasting >30 Seconds at the Last Follow-up Visit in the Absence of Class I or III AADs.
Description: Freedom from any documented AF, AFL, or AT lasting >30 seconds at the last follow-up visit in the absence of Class I or III AADs.
Time Frame: 12-24 months post procedure
Reporting Status: Not Posted

5. Secondary Outcome: Acute Procedural Success Defined as Documentation of Sinus Rhythm at the End of the Procedure.
Description: Acute procedural success defined as documentation of sinus rhythm at the end of the procedure.
Time Frame: At end of procedure
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Freedom From Pacemaker Implant or Overall Device or Surgical Ablation Procedures Related to Adverse Events
Description: Freedom from pacemaker implant or overall device or Surgical Ablation procedures Related to Adverse Events
Time Frame: 12-24 months post procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: At time of procedure
Arm/Group | Non-Randomized, Single Arm Study
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 12/33
Other Adverse Events (participants affected / at risk) | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Randomized, Single Arm Study (N=33)
Complete Heart Block (Cardiac disorders) | 2
Aneurysm (Cardiac disorders) | 1
Atrioventricular Block (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Sick Sinus Syndrome (Cardiac disorders) | 1
Other (Cardiac disorders) | 2
Other (Metabolism and nutrition disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT05089877/Prot_SAP_000.pdf